CLINICAL TRIAL: NCT03157037
Title: Open-Label Phase II Study in Anti-GBM Disease (Goodpasture's Disease) With Adverse Renal Prognosis to Evaluate the Efficacy and Safety of IdeS - GOOD-IDES
Brief Title: Open-Label Phase II Study to Evaluate the Efficacy and Safety of IdeS in Anti-GBM Disease
Acronym: GOOD-IDES-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mårten Segelmark (Other Government)
Collaborators: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor-Investigator, Mårten Segelmark, MD, PhD and Professor Department of Drug Research, Department of Medical and Health Sciences, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOOD-IDES-01
Record Dates: First submitted 2017-05-11; First posted 2017-05-17 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Anti-Glomerular Basement Membrane Antibody Disease
MeSH Terms: conditions — Rapidly progressive glomerulonephritis with pulmonary hemorrhage | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Intervention Model Description: Open-Label, Single Arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imlifidase (Experimental): Imlifidase 0.25 mg/kg body weight intravenous infusion
  Interventions: Biological: Imlifidase

INTERVENTIONS:
Biological: Imlifidase — One dose of 0.25 mg/kg body weight imlifidase on study day 1
  Other Names: Immunoglobulin G-degrading enzyme of Streptococcus pyogenes; HMed-IdeS; IdeS

SUMMARY:
This study will evaluate the safety and tolerability of IdeS in patients with severe anti-glomerular basement membrane (anti-GBM) disease receiving standard of care consisting of pulse-methylprednisolone, oral prednisolone and intravenous cyclophosphamide combined with plasma exchange (PLEX).

DETAILED DESCRIPTION:
This is an Open-Label Phase 2 Study to Evaluate the Efficacy and Safety of IdeS in anti-GBM disease (Goodpasture's disease, i.e. GP) with Adverse Renal Prognosis. The primary efficacy objective is to evaluate the efficacy of an IdeS based regimen to salvage independent renal function measured as no need for dialysis at 6 months after IdeS treatment. The primary safety objective of this study is to evaluate the safety and tolerability of IdeS in patients with severe anti-GBM disease on background of standard care consisting of pulse-methylprednisolone, oral prednisolone and intravenous cyclophosphamide (CYC) combined with plasma exchange (PLEX). The patients will be followed during 6 months according to the study visit plan.

ELIGIBILITY:
Inclusion Criteria:

1. Anti-GBM antibodies detected by ELISA above a level that is considered toxic by the investigator using local laboratory. Patients double-positive for anti-GBM and anti-neutrophil cytoplasmic antibodies (ANCAs) may be entered in the trial, but only if their level of anti-GBM antibodies fulfil the criteria listed above.
2. Estimated glomerular filtration rate (eGFR) <15 ml/min/1.73 m^2 (by modification of diet in renal disease (MDRD) equation) or if the patient is non-responsive to standard treatment, and has lost >15 ml/min/1.73 m^2 after start of treatment
3. Haematuria on dipstick and/or urinary sediment
4. Male or female patients aged at least 18 years; Female patients of childbearing potential may participate if highly effective contraception is used during the study, according to Clinical Trials Facilitation and Coordination Group (CTFG) guidance [18], see also section 4.9 (pregnancy test should be performed before inclusion).
5. Willing and able to give written Informed Consent and to comply with the requirements of the study protocol; and
6. Judged to be otherwise healthy by the Investigator, based on medical history, physical examination, and clinical laboratory assessments. Patients with clinical laboratory values that are outside of normal limits (other than those specified in the Exclusion Criteria) and/or with other abnormal clinical findings that are judged by the Investigator not to be of clinical significance, may be entered into the study.

Exclusion Criteria:

1. Anuria for more than 2 days (less than 200 ml during last 48 hours);
2. Dialysis dependency for more than 5 days (maximum 3 sessions before signing informed consent);
3. Ongoing moderate to severe pulmonary haemorrhage (or having ceased within the last two weeks), defined as requiring assisted ventilation, oxygen or blood transfusions.
4. Pregnancy.
5. Symptomatic congestive heart failure (NYHA class 2-4) and requiring prescription medication or clinically evident peripheral edema of cardiac origin;
6. Myocardial infarction, unstable angina or stroke within 3 months prior to screening;
7. Ongoing bacterial infection requiring antibiotic therapy or viral infection with Hepatitis B, C or HIV (up to 3 months old negative test results are accepted); or active tuberculosis as indicated by chest x-ray.
8. Patients should not have received investigational drugs within 30 days prior to screening or within 4 half-lives (whichever is longer); and
9. History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the subject at unacceptable risk for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Segelmark, MD PhD Prof, Principal Investigator — Linkoeping University
Locations (10):
- Department of Internal Medicine IV (Nephrology and Hypertension), Innsbruck, Austria
- Department of Department of nephrology, First Faculty of Medicine and General Teaching Hospital and Charles University in Prague, Czech Republic,, Prague, Czechia
- Department of Department of Nephrology, Rigshospitalet, Copenhagen, Copenhagen, Denmark
- France (5):
  - PH USI UNTR, service du Pr Rondeau, Hôpital Tenon, Paris, Paris Cedex 20
  - Department of Nephrology, Hemodialysis, Apheresis, and Transplantation, CHUGA (centre hospitalier universitaire Grenoble-Alpes), Grenoble
  - Centre Hospitalier Régional Universitaire de Lille, Nephrology Service, Lille
  - Nephrology Service CHU Bichat, Paris
  - Department of Nephrology and Organ Transplant, CHU Rangueil, Toulouse
- Sweden (2):
  - Karolinska University Hospital Huddinge, Stockholm
  - Department of Nephrology, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berden AE, Ferrario F, Hagen EC, Jayne DR, Jennette JC, Joh K, Neumann I, Noel LH, Pusey CD, Waldherr R, Bruijn JA, Bajema IM. Histopathologic classification of ANCA-associated glomerulonephritis. J Am Soc Nephrol. 2010 Oct;21(10):1628-36. doi: 10.1681/ASN.2010050477. Epub 2010 Jul 8. PMID 20616173
- [Background] van Daalen EE, Jennette JC, McAdoo SP, Pusey CD, Alba MA, Poulton CJ, Wolterbeek R, Nguyen TQ, Goldschmeding R, Alchi B, Griffiths M, de Zoysa JR, Vincent B, Bruijn JA, Bajema IM. Predicting Outcome in Patients with Anti-GBM Glomerulonephritis. Clin J Am Soc Nephrol. 2018 Jan 6;13(1):63-72. doi: 10.2215/CJN.04290417. Epub 2017 Nov 21. PMID 29162595
- [Derived] Tyrberg L, Andersson F, Uhlin F, Hellmark T, Segelmark M. Using imlifidase to elucidate the characteristics and importance of anti-GBM antibodies produced after start of treatment. Nephrol Dial Transplant. 2023 Dec 20;39(1):45-54. doi: 10.1093/ndt/gfad132. PMID 37385828

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment HMed-IdeS: A single dose of IdeS (imlifidase) 0.25 mg/kg body weight (BW) intravenous infusion on study Day 1
Period: Overall Study
Arm/Group | Treatment HMed-IdeS
Started | 15
Completed | 14
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Imlifidase: IdeS intravenous infusion 0.25 mg/kg body weight (BW) intravenous infusion
  HMed-IdeS: One dose of 0.25 mg/kg BW HMed-IdeS on study day 1
Arm/Group | Imlifidase
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 61 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 4
  Austria | 2
  Czechia | 1
  Denmark | 3
  France | 5
Dialysis status at baseline [Count of Participants; unit: Participants]
  Dialysis | 10
  Not on dialysis but eGFR <15 mL/min/1.73 m^2 | 5
Time since anti-glomerular basement membrane (anti-GBM) diagnosis [Median (Full Range); unit: days] | 2 [0 to 40]
Anti-GBM concentration [Median (Full Range); unit: U/mL] | 130 [2 to 1090]
Time since first renal symptom [Median (Full Range); unit: days] | 10 [4 to 76]
Occurrence of pulmonary symptom [Count of Participants; unit: Participants]
  Yes | 9
  No | 3
  Not reported | 3
Time since first pulmonary symptom [Median (Full Range); unit: days] | 32 [1 to 113]
Double positive Anti-GBM and antineutrophil cytoplasmic antibodies (ANCA) [Count of Participants; unit: Participants] — ANCA=anti-neutrophil cytoplasm antibody
  Participants
    Yes | 6
    No | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Independent Renal Function at 6 Months
Description: Number of patients without need for dialysis at 6 months. A patient with independent renal function is defined as a patient without need for dialysis.
Time Frame: 6 months after dosing
Measure: Count of Participants; unit: Participants
Groups:
- Dialysis Dependent at Baseline: Patients who were dialysis dependent at baseline
- Dialysis Independent at Baseline: Patients who were dialysis independent at baseline
- All Patients: All patients (i.e., both patients who were dialysis dependent and patients who were dialysis independent at baseline)
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 10 | 5 | 15
Participants | 5 | 5 | 10

2. Secondary Outcome: Number of Patients With Independent Renal Function at 3 Months
Description: Number of patients without need for dialysis at 3 months. A patient with independent renal function is defined as a patient without need for dialysis.
Time Frame: 3 months after dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 10 | 5 | 15
Participants | 4 | 5 | 9

3. Secondary Outcome: Renal Function at 3 and 6 Months
Description: Estimated glomerular filtration rate (eGFR) is a measure of kidney function. eGFR was calculated based on p-creatinine according to the modification of diet in renal disease (MDRD) equation.
  eGFR for a kidney with normal function is above 90 mL/min/1.73m^2. Reduced kidney function is characterised by a decreased eGFR value.
Time Frame: 3 and 6 months after imlifidase dosing
Population: Only patients who were alive and dialysis independent at respective analysis time (3 and 6 months) were included in this analysis because assessment of eGFR is not considered meaningful for patients in dialysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 5 | 5 | 10
mL/min/1.73m^2
  eGFR at 3 months: number analyzed (Participants) | 3 | 4 | 7
  eGFR at 3 months | 20.3 (4.7) | 26.5 (11.0) | 23.8 (8.9)
  eGFR at 6 months | 24.8 (6.6) | 36.9 (17.3) | 30.9 (13.9)

4. Secondary Outcome: Number of Patients With Renal Function Over Time Stratified by Ranges of eGFR
Description: eGFR is a measure of kidney function. eGFR has been calculated based on p-creatinine according to the modification of diet in renal disease (MDRD) equation.
  eGFR for a kidney with normal function is above 90 mL/min/1.73m^2. Reduced kidney function is characterised by a decreased eGFR value.
  Number of patients per 4 different eGFR categories (0-15, 15-30, 30-60, ≥60 mL/min/1.73m^2) are presented. A shift towards a higher category during the study indicates improved renal function over time.
Time Frame: Pre-imlifidase, 1, 3 and 6 months after imlifidase dosing
Population: Only patients who were alive and dialysis independent at each specific analysis time are included in this analysis because eGFR is not applicable for patients in dialysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 5 | 5 | 10
Participants
  Pre-imlifidase: number analyzed (Participants) | 1 | 5 | 6
  Pre-imlifidase: eGFR (0-15) | 1 | 5 | 6
  Pre-imlifidase: eGFR (15-30) | 0 | 0 | 0
  Pre-imlifidase: eGFR (30-60) | 0 | 0 | 0
  Pre-imlifidase: eGFR (≥60) | 0 | 0 | 0
  Month 1: number analyzed (Participants) | 2 | 5 | 7
  Month 1: eGFR (0-15) | 1 | 1 | 2
  Month 1: eGFR (15-30) | 1 | 2 | 3
  Month 1: eGFR (30-60) | 0 | 2 | 2
  Month 1: eGFR (≥60) | 0 | 0 | 0
  Month 3: number analyzed (Participants) | 3 | 4 | 7
  Month 3: eGFR (0-15) | 0 | 0 | 0
  Month 3: eGFR (15-30) | 3 | 3 | 6
  Month 3: eGFR (30-60) | 0 | 1 | 1
  Month 3: eGFR (≥60) | 0 | 0 | 0
  Month 6: eGFR (0-15) | 0 | 0 | 0
  Month 6: eGFR (15-30) | 4 | 2 | 6
  Month 6: eGFR (30-60) | 1 | 3 | 4
  Month 6: eGFR (≥60) | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Anti-GBM Antibodies Above a Toxic Level Stratified by Number of Study Visits
Description: Anti-GBM antibodies above a toxic level defined as >20 U/mL. The level of anti-GBM antibodies was measured centrally using the Phadia ELiA(TM) anti-GBM kit. The enzyme-linked immunoassay (ELiA) is a fluorescence enzyme immunoassay.
Time Frame: Predose up to 6 months after dosing
Population: Number of study visits with a toxic level are presented instead of number of patient days with an anti-GBM level >20 U/mL as was the original plan.
Measure: Number; unit: participants
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 10 | 5 | 15
participants
  0 visits | 1 | 1 | 2
  1 visit | 3 | 4 | 7
  2 visits | 1 | 0 | 1
  3 visits | 1 | 0 | 1
  5 visits | 2 | 0 | 2
  6 visits | 1 | 0 | 1
  9 visits | 1 | 0 | 1

6. Secondary Outcome: Number of Patients With Haematuria (Blood in Urine)
Description: Haematuria was assessed using urine dipstick. The result was presented as: Negative/Trace/+1/+2/+3/+4.
  In the analysis results being +2 or above are considered as relevant. Haematuria was an inclusion criterion. All 15 patients had haematuria when included in the study.
Time Frame: At 6 months after dosing
Population: Data was missing for 5 of the 15 patients at 6 months.
Measure: Number; unit: Patients with haematuria (+2 or above)
Arm/Group | All Patients
Number analyzed (Participants) | 10
Patients with haematuria (+2 or above) | 3

7. Secondary Outcome: Change in Proteinuria During the Study
Description: Change in proteinuria measured as u-albumin/creatinine (g/mol) in morning void during the study .
Time Frame: Pre-imlifidase, 3 and 6 months after imlifidase dosing
Population: Some patients had missing data at some visits
Measure: Mean (Standard Deviation); unit: g/mol
Groups:
- All Patients: All patients irrespective of dialysis dependency at baseline and at 6 months
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 10 | 5 | 15
g/mol
  Pre-imlifidase: number analyzed (Participants) | 6 | 5 | 11
  Pre-imlifidase | 1117 (1544) | 199 (166) | 700 (1197)
  3 months: number analyzed (Participants) | 5 | 4 | 9
  3 months | 220 (197) | 153 (172) | 190 (178)
  6 months: number analyzed (Participants) | 9 | 5 | 14
  6 months | 183 (231) | 122 (133) | 161 (198)

8. Secondary Outcome: Number of PLEXs Needed Over Time
Description: Number of PLEXs needed before anti-GBM antibodies are below toxic levels. PLEX was initiated at the discretion of the investigator throughout the study.
Time Frame: Pre-screening and up to Day 93 after imlifidase dosing
Measure: Number; unit: Number of PLEX performed
Groups:
- All Patients: All patients irrespective of dialysis dependency at baseline
Arm/Group | Dialysis Dependent at Baseline | Dialysis Independent at Baseline | All Patients
Number analyzed (Participants) | 10 | 5 | 15
Number of PLEX performed
  Pre-Screening | 10 | 23 | 33
  Post-Screening to pre-imlifidase dose | 5 | 0 | 5
  Pre-imlifidase to Day 3 | 0 | 1 | 1
  Day 3 to Day 7 | 8 | 0 | 8
  Day 7 to Day 10 | 14 | 0 | 14
  Day 10 to Day 15 | 20 | 2 | 22
  Day 15 to Day 22 | 18 | 5 | 23
  Day 22 to Day 29 | 5 | 1 | 6
  Day 29 to Day 50 | 5 | 3 | 8
  Day 50 to Day 93 | 0 | 1 | 1
  Total (post-imlifidase to Day 93) | 70 | 13 | 83
  Total (pre-screening to Day 93) | 85 | 36 | 121

9. Secondary Outcome: Pharmacokinetics of Imlifidase (Cmax)
Description: Maximum observed plasma concentration of IdeS following dosing (Cmax)
Time Frame: Pre-dose, 45min, 2h, 6h, 24h, Day3, Day 7, Day 10, and Day15
Measure: Geometric Mean (Full Range); unit: µg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 15
µg/mL | 4.7 [2.6 to 8.0]

10. Secondary Outcome: Pharmacokinetics of Imlifidase (AUC)
Description: Area under the plasma concentration versus time curve (AUC)
Time Frame: Pre-dose, 45min, 2h, 6h, 24h, Day3, Day 7, Day 10, and Day15
Measure: Geometric Mean (Full Range); unit: h*µg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 15
h*µg/mL | 158 [73 to 304]

11. Secondary Outcome: Pharmacokinetics of Imlifidase (t1/2)
Description: Half-life during distribution phase (Alpha-t1/2) Half-life during elimination phase (Beta-t1/2) The results refers to harmonic mean.
Time Frame: Pre-dose, 45min, 2h, 6h, 24h, Day3, Day 7, Day 10, and Day15
Measure: Mean (Full Range); unit: h
Arm/Group | All Patients
Number analyzed (Participants) | 15
h
  Alpha-t1/2 | 2.6 [0.9 to 7.5]
  Beta-t1/2 | 53 [26 to 115]

12. Secondary Outcome: Pharmacokinetics of Imlifidase (CL)
Description: Clearance (CL) is a measure of the ability of the body to clear imlifidase from plasma
Time Frame: Pre-dose, 45min, 2h, 6h, 24h, Day3, Day 7, Day 10, and Day15
Measure: Geometric Mean (Full Range); unit: mL/h/kg
Arm/Group | All Patients
Number analyzed (Participants) | 15
mL/h/kg | 1.6 [0.8 to 3.4]

13. Secondary Outcome: Pharmacokinetics of Imlifidase (Vz)
Description: Vz = Volume of distribution during the elimination phase
Time Frame: Pre-dose, 45min, 2h, 6h, 24h, Day3, Day 7, Day 10, and Day15
Measure: Geometric Mean (Full Range); unit: L/kg
Arm/Group | All Patients
Number analyzed (Participants) | 15
L/kg | 0.13 [0.07 to 0.21]

14. Secondary Outcome: Pharmacodynamics (IgG Degradation Measured as Remaining Concentration of Intact and Single Cleaved IgG)
Description: Imlifidase specifically cleaves all subclasses of human IgG rapidly and efficiently.
  The cleaving process involves two steps: (i) intact IgG to single cleaved IgG followed by (ii) single cleaved IgG to completely cleaved IgG (one F(ab')2- and one homodimeric Fc-fragment) The electroluminescence analysis method used measures the sum of intact and single cleaved IgG in serum.
  The efficacy of imlifidase is evaluated as remaining concentration of intact and single cleaved IgG in serum after treatment.
Time Frame: Pre-dose up to 6 months after imlifidase administration
Population: Some patients had missing data at some timepoints
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 15
mg/mL
  Pre-dose | 6.66 (2.94)
  2 hours | 0.17 (0.12)
  6 hours | 0.08 (0.05)
  24 hours: number analyzed (Participants) | 14
  24 hours | 0.08 (0.05)
  Day 3 | 0.09 (0.05)
  Day 7 | 0.85 (1.56)
  Day 10 | 1.58 (1.69)
  Day 15 | 2.64 (2.42)
  Day 22 | 2.94 (2.34)
  Day 29 | 3.94 (2.18)
  Day 50: number analyzed (Participants) | 14
  Day 50 | 4.29 (2.05)
  Day 180: number analyzed (Participants) | 14
  Day 180 | 6.76 (2.49)

15. Secondary Outcome: Anti-imlifidase Antibodies (ADA)
Description: Determination of anti-imlifidase antibody concentration
Time Frame: Up to 6 months after dosing
Population: Some missing data at Day 50, Day 93 and Day 180
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- All Patients: All patients (i.e., irrespective of dialysis dependency at baseline)
Arm/Group | All Patients
Number analyzed (Participants) | 15
mg/L
  Pre-imlifidase | 9.00 (4.17)
  Day 7 | 4.32 (5.29)
  Day 15 | 752 (728)
  Day 22 | 744 (736)
  Day 29 | 609 (493)
  Day 50: number analyzed (Participants) | 14
  Day 50 | 547 (580)
  Day 93: number analyzed (Participants) | 12
  Day 93 | 327 (263)
  Day 180: number analyzed (Participants) | 14
  Day 180 | 242 (280)

16. Secondary Outcome: Renal Histology
Description: Kidney biopsies were classified according to the histopathologic classification for antineutrophil cytoplasmic antibodies (ANCA)-associated glomerulonephritis developed by Berden et al. 2010.
  This classification has previously been applied in a study of 123 anti-GBM disease patients (von Daalen et al 2018).
  Histopathologic class:
  * Focal (≤50% normal glomeruli)
  * Crescentic (≥50% glomeruli with cellular crescents)
  * Mixed (<50% normal, <50%crescentic, <50% globally sclerotic glomeruli)
  * Sclerotic (≥50% globally sclerotic glomeruli) In addition information on the histological activity and kidney outcome was provided.
  Focal class is associated with favourable kidney outcome, whereas sclerotic carries a poor outcome. Crescentic/mixed class could have an intermediate outcome between focal and sclerotic.
  Immunofluorescence performed at the local hospitals was also used to assess linear IgG deposits which is a hallmark of anti-GBM antibody disease.
Time Frame: Before administration of imlifidase (0-33 days) and after administration of imlifidase (3-6 days)
Population: During the study, 14 kidney biopsies were taken from 10 of the 15 included patients. 10 biopsies were taken before administration of imlifidase and 4 after administration of imlifidase.
Measure: Number; unit: Biopsies
Units Other Than Participants: Biopsies
Groups:
- 14 Biopsies Collected From 10 Patients in the Study: 10 biopsies were collected before imlifidase administration and 4 biopsies were collected after imlifidase administration
Arm/Group | 14 Biopsies Collected From 10 Patients in the Study
Number analyzed (Participants) | 10
Number analyzed (Biopsies) | 14
Biopsies
  Crescentic | 9
  Mixed | 4
  Sclerotic | 1
  Linear IgG deposits | 11

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 6 months (i.e., from the timepoint the patient signed the informed consent form (ICF) until end of study. A treatment emergent adverse event (TEAE) is defined as any AE occurring after imlifidase administration and within the time of the residual drug effect period (i.e. 28 days after admin).
Description: Data on AEs were obtained if spontaneously reported, if reported in response to an open question, or if revealed by observation.
  All Serious Adverse Events (SAEs) were post-TEAEs and those are listed in the "SAE" table.
  "Other (Not Including Serious) Adverse Events" presents all reported AEs in the study (47 TEAEs and 35 post-TEAEs).
Groups:
- Safety Analysis Set: All patients who have received imlifidase.
Arm/Group | Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=15)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=15)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 2 (3)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Cryoglobulinaemia (Immune system disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Blood iron decreased (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Anti-glomerular basement membrane antibody positive (Investigations) | 1 (1)
Borrelia test positive (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT03157037/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03157037/SAP_001.pdf